CLINICAL TRIAL: NCT05051761
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of Jaktinib in Adult Patients With Severe Alopecia Areata
Brief Title: Study to Evaluate the Safety and Efficacy of Jaktinib in Adults With Alopecia Areata
Acronym: AA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZGJAK018
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib 50mg BID (Experimental): Participants received Jaktinib 50mg tablets, orally, twice daily (BID) for up to 24 weeks.
  Interventions: Drug: Jaktinib
- Jaktinib 75mg BID (Experimental): Participants received Jaktinib 75mg tablets, orally, twice daily (BID) for up to 24 weeks.
  Interventions: Drug: Jaktinib
- placebo (Placebo Comparator): Participants received Jaktinib matched placebo tablets, orally, twice daily (BID) for up to 24 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Jaktinib — Administered orally.
  Arms: Jaktinib 50mg BID; Jaktinib 75mg BID
Drug: placebo — Administered orally.
  Arms: placebo

SUMMARY:
This is a multi-center Phase 3 study to evaluate the safety and effectiveness of an investigational study drug (called Jaktinib) in adults (≥18 years and <65 years) who have 50% or greater scalp hair loss. The study is placebo-controlled, meaning that some patients entering the study will not receive active study drug but will receive tablets with no active ingredients (a placebo). It is double-blinded, meaning that the Sponsor, the study doctors, the staff, and the patients will not know whether a patient is on active study drug (or the dose) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* participants voluntarily sign the informed consent form (ICF);
* Age ≥ 18 years and <65 years, either male or female;
* Clinical presentation compatible with alopecia areata with a current episode lasting not exceeding ≤8 years.
* At least 50% scalp hair loss.
* Willing to comply with the study visits and requirements of the study protocol.

Exclusion Criteria:

* participants has taken a JAK inhibitor prior to randomization;
* participants who are unsuitable to the trial, as identified by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Severity of Alopecia Tool (SALT) ≤ 20 at Week 24 | Week 24
  SALT is a quantitative assessment of scalp hair loss with scores ranging in severity from 0 (no scalp hair loss) to a maximum of 100 (complete scalp hair loss).

SECONDARY OUTCOMES:
Percentage of Participants Achieving 50% Improvement of SALT (SALT50) | Week 24
  Percentage of participants achieving SALT50

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Hospital for Skin Diseases, Chinese Academy of medical Sciences, Nanjing, Jiangsu